CLINICAL TRIAL: NCT07209813
Title: A Phase Ⅱ, Multicenter, Parallel Comparison Clinical Study of GKL-006 Combined With TACE in Treatment of Unresectable Hepatocellular Carcinoma
Brief Title: GKL-006 Combined With TACE in Treatment of Unresectable Hepatocellular Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Gene Key Life Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023LP02333
Record Dates: First submitted 2025-09-29; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GKL-006 (Experimental): Experimental group: GKL-006（3.0±0.9）×108 iNKT cells/m2)+TACE
  Interventions: Biological: GKL-006
- TACE (Active Comparator): TACE
  Interventions: Biological: GKL-006

INTERVENTIONS:
Biological: GKL-006 — GKL-006（3.0±0.9）×108 iNKT cells/m2 IV single infusion on Day 1 of each 14-day cycle for up to 11 cycles (≈6 month) in the absence of disease progression or unacceptable toxicity.

SUMMARY:
This is a Phase II, open-label, randomized, multicenter study to evaluate the efficacy and safety of GKL-006 combine with TACE in adult patients with unresectable Hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* 1.Be willing and able to provide written informed consent/assent for the trial 2.Male or female, ≥ 18 years of age, ≤ 75 years of age. 3.Hepatocellular carcinoma confirmed as unresectable by histopathology/cytology/imaging studies (such as dynamic CT or MRI) 4. With a total tumor volume not exceeding 50% of the liver, a maximum diameter of a single tumor not exceeding 7 cm, and a total number of target lesions and non-target lesions not exceeding 10 5.Patients must have at least one measurable lesion by mRECIST criteria. 6.Have an overall Child-Pugh score ≤9 7.Have a performance status of 0 to 2 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale 8.Have life expectancy of ≥ 6 months. 9.The subject has adequate hematological and organ function, and the laboratory test results within 14 days before randomization

Exclusion Criteria:

* 1.Subjects with a history of (within 5 years) or concurrent other untreated malignant tumors, except for cured basal cell carcinoma of the skin, carcinoma in situ, and breast cancer that has been recurrence-free for more than 3 years after completing radical resection.

  2.Have previous organ transplantation 3.Known fibrolamellar HCC or mixed hepato-cholangiocarcinoma. 4. Patients receive radiotherapy within the 4 weeks preceding study enrolment;Patients receive Chinese traditional medicine for cancer treatment within the 2 weeks preceding study enrolment; 5. Patients must not have had any surgical procedure requiring hospitalization and administration of general anesthesia within the past 4 weeks.

  6. Patients with autoimmune disease. 7.Have serious illnesses including, but not limited to, congestive heart failure (NYHA class III or IV functional classification);Left Ventricular Ejection Fraction (LVEF) < 50% on echocardiogram;life threatening cardiac arrhythmia; or myocardial infarction or cerebral vascular accident within the last 6 months.

  8. Uncontrolled high blood pressure (systolic blood pressure, SBP ≥140 mmHg and/or diastolic blood pressure, DBP ≥90 mmHg).

  9. Has a known history of Human Immunodeficiency Virus (HIV,Syphilis,or other). 10. Pregnant or breast-feeding. 11. Has received a live vaccine within the 4 weeks preceding study enrolment; 12. Has participated in other clinical studies within the 4 weeks preceding study enrolment; 13. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating Principal Investigator (PI).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 48 (Estimated)
Dates: Start 2025-10-12 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | From enrollment to the end of treatment at 6 month